CLINICAL TRIAL: NCT06423885
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-M07D1 Combination Therapy in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of BL-M07D1 Combination Therapy in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-206
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received BL-M07D1+PD-1 monoclonal antibody in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-M07D1; Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: PD-1 monoclonal antibody — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a multicenter, open-label, phase II clinical study to explore the safety and efficacy of BL-M07D1+PD-1 monoclonal antibody in patients with unresectable locally advanced or metastatic HER2-positive gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age ≥18 years old and ≤75 years old at the time of signing the informed consent;
4. Expected survival time ≥3 months;
5. Patients with HER2-positive gastric or gastroesophageal junction adenocarcinoma confirmed by pathology;
6. Patients provided tumor tissue specimens as far as possible for the detection of biomarkers such as HER2 and PD-L1 for exploratory retrospective analysis;
7. Must have at least one measurable lesion according to RECIST v1.1 definition;
8. ECOG 0 or 1;
9. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. Blood transfusion is not allowed within 14 days before the first use of study drugs, and the use of colony-stimulating factors is not allowed, and the organ function level must meet the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN;
13. Urine protein ≤2+ or ≤1000mg/24h;
14. Female subjects of childbearing potential, or male subjects with a fertile partner, had to use highly effective contraception from 7 days before the first dose until 7 months after the dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Anti-tumor therapy such as chemotherapy, biological therapy, and immunotherapy had been used within 4 weeks or 5 half-lives before the first dose. Oral drugs such as fluorouracil;
2. Prior ADC drug therapy with camptothecin derivative as toxin;
3. The history of severe cardiovascular and cerebrovascular diseases in the past six months;
4. Serious impairment of lung function due to pulmonary diseases;
5. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
6. Other primary malignancies diagnosed within 5 years before the first dose;
7. Poorly controlled hypertension;
8. A history of ILD requiring steroid therapy, current ILD/interstitial pneumonia or suspected to have such a condition during screening;
9. Patients with active central nervous system metastases;
10. Patients who are allergic to any excipients of the trial drug;
11. Systemic corticosteroids or immunosuppressive agents are required within 2 weeks before study dosing;
12. Patients with massive or symptomatic effusions or poorly controlled effusions;
13. Severe systemic infection within 4 weeks before screening;
14. Active autoimmune and inflammatory diseases;
15. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
16. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
17. A history of severe neurological or psychiatric illness;
18. Pregnant or lactating women;
19. The presence of other serious physical or laboratory abnormalities or poor compliance may increase the risk of participating in the study risk, or interference with the results of the study, and patients who were deemed by the investigators to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M07D1 to the first date of either disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  he DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China